CLINICAL TRIAL: NCT03969082
Title: Bibliotherapy, Students in Medicine and Health Sciences Read to Patients With Cancer During Treatment, an Evaluation by Patients and Students.
Brief Title: Evaluation of Bibliotherapy by Students and Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other); Het Lezerscollectief (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BC-4703
Record Dates: First submitted 2019-04-24; First posted 2019-05-31 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Acute Leukemia; Advanced Solid Tumor
Keywords: Bibliotherapy; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Bibliotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bibliotherapy (Experimental): Students will read to patients receiving active treatment using the "read aloud" method. This will be performed in a 1: 1 relationship for half an hour for 8-10 times during a period of six months.
  Interventions: Behavioral: Bibliotherapy

INTERVENTIONS:
Behavioral: Bibliotherapy — Students will read to patients during 30 minutes. They will read aloud and pause regularly to encourage patients to reflect on what is being read, on the thoughts the poem or book has stirred or on how the reading matter relates to their own lives.

SUMMARY:
Research has demonstrated the positive effects of bibliotherapy (the use of reading in the treatment of patients), such as increased self-awareness, increased empathy, hope and decreased negativity. At Ghent University Hospital, 20 students from the Faculty of Medicine and Health Sciences were selected to be trained as readers by 'The Readers Collective', a Flemish Organization inspired by The Reader. Those students will read to patients with acute leukemia or to patients with a solid tumors in an advanced stage, using the "read aloud" method. Eight to ten reading sessions of approximately half an hour will be organized in a 1: 1 relationship between student and patient during a period of six months. The primary aim of study is to determine the acceptability and feasibility of the intervention by the patients as well as the students. Secondary aims are exploring the impact of the reading sessions on the professional development of the students and on the emotional well-being and quality of life of cancer patients. Assessment will be based upon questionnaires (as a basis for the in-depth interviews), diary notes, and in-depth interviews.

DETAILED DESCRIPTION:
Bibliotherapy has been defined in different ways, but fundamentally means helping people through the use of books. In clinical contexts, it often refers to psychological self-help interventions that use treatment books [1]. However, other reading therapies exist, such as reading to patients during their treatment. Studies have demonstrated the positive effects of the use of reading in the treatment of patients such as increased self-awareness, empathy and hope and less negativity. The Reader, a British national charity, is the pioneer of a specific literature-based intervention i.e. shared reading. This approach is different from many reading therapies because it emphasizes on (1) reading aloud so that the book is a live presence and not an object of study (as is the case in educational settings) or a subject of chat (as in a book club) and on (2) literature (poetry and fiction) and its role in offering a model of human thinking and feeling. In the model of The Reader, small groups (2-12 people) come together weekly, to read novels, short stories and poetry together aloud. The target groups of The Reader are very diverse such as ordinary library visitors, vulnerable youth, rehabilitation groups in psychiatric hospitals, groups in prisons, prevention groups for stress and burnout, growth groups, personal etc.

This project, however, is unique in different ways. First, reading sessions will be organized in the hospital setting in a 1:1 relationship, as opposed to in small groups. Second, we will asses the possible impact of the intervention on emotional wellbeing and quality of life of patients with cancer, as well as on the student's professional development. This will be done by means of questionnaires (not as a quantitative study, but as a basis for the in-depth interview), diary notes, and an in-depth interview (student and patient separately and once together) .

The primary aim of this project is to assess the acceptability of this intervention. Specifically, this study seeks feedback on how well the reading sessions are received by the patients and the students. Secondly, we will assess if the sessions meet the needs of patients in their coping with cancer and help students in their professional development. To assess acceptability, in-depth interviews will be used and participants will be asked about their opinions regarding the reading sessions. We chose this particular interview type because it grants the interviewer flexibility to follow up with relevant questions and probes to gather richer information. The interviews will be recorded for transcription and analysis.

A call for participation for this study was made to students in Medicine and Health Sciences of Ghent University at a lecture of Jane Davis, the founder of The Reader. Students could submit their application; in total more than 50 applications were received. Three physicians (Dr. Helewaut, Dr. Pype and Dr. Kerre) independently scored the applications on the basis of motivation, background and age.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Clinical diagnosis of acute leukemia or advanced cancer of a solid tumor
* Treated at an inpatient ward (for patients with leukemia)
* Treated at inpatient ward ( for patients with solid tumor)

Exclusion Criteria:

* Patients under 18 years;
* Patients who are not able to read or understand Dutch.

Students:

- Student of the Faculty of Medicine and Health Sciences of Ghent University

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention | Interviews after six months of the first reading session
  In-depth interview will be used to seek feedback on how well the reading session are received by the patients and the students

SECONDARY OUTCOMES:
Impact of the intervention | Questionnaires: baseline, 12 weeks and six months;
  Impact on Quality of Life measured by the European Organisation for Research and Treatment of Cancer Quality of Life C30 questionnaire, score range 0-100, 100 is better score
Impact of intervention in student by the use of in-depth interviews | In-depth interviews at 12 weeks and after six months of the first reading session
  Impact on professional development of students in Medicine and Health Sciences by performing in-depth interviews
Acceptability of the intervention | Interviews after 3 months of the first reading session
  In-depth interview will be used to seek feedback on how well the reading session are received by the patients and the students
Effect on quality of life of patients | Questionnaires: baseline, 12 weeks and six months
  Effect of quality of life with the McGill Quality of Life Scale, range 0-10, higher score is better score
Effect on mood of patients | Questionnaires: baseline, 12 weeks and six months
  Hospital Anxiety and Depression Scale, range 0-21, higher score is worse score
Effect on depression of patients | Questionnaires: baseline, 12 weeks and six months
  Patient Health Questionnaire-9, range 0-27, higher score is worse score

OTHER OUTCOMES:
Feasibility of the intervention: Feedback based upon in-depth interviews organised | Interviews at 12 weeks after the first reading session
  Feedback based upon in-depth interviews organised
Feasibility of the intervention by looking at number of reading sessions per dyad | Six months
  Number of reading sessions organized
Feasibility of the intervention measured with in-depth interviews | Interviews after six months of the first reading session
  Feedback based upon in-depth interviews organised

CONTACTS AND LOCATIONS:
Overall Officials: Tessa Kerre, PhD, Principal Investigator — Department of Hematology, Ghent University Hospital; Vibbeke Kruse, PhD, Study Chair — Department of Medical Oncology/ Cancer Center, Ghent University Hospital; Peter Pype, PhD, Study Chair — Department of Public Health and Primary Care, Ghent University; Fleur Helewaut, Study Chair — Clinical Skills Training Centre, Ghent University; Jan Raes, Study Chair — Founder, Het Lezerscollectief
Locations (1):
- Universitair Ziekenhuis Gent, Ghent, Oost-Vlaanderen, Belgium

REFERENCES:
- [Background] Malibiran R, Tariman JD, Amer K. Bibliotherapy: Appraisal of Evidence for Patients Diagnosed With Cancer. Clin J Oncol Nurs. 2018 Aug 1;22(4):377-380. doi: 10.1188/18.CJON.377-380. PMID 30035795
- [Background] Davis J. Enjoying and enduring: groups reading aloud for wellbeing. Lancet. 2009 Feb 28;373(9665):714-5. doi: 10.1016/s0140-6736(09)60426-8. No abstract available. PMID 19263586
- [Result] Korner A, Roberts N, Steele RJ, Brosseau DC, Rosberger Z. A randomized controlled trial assessing the efficacy of a self-administered psycho-educational intervention for patients with cancer. Patient Educ Couns. 2019 Apr;102(4):735-741. doi: 10.1016/j.pec.2018.12.002. Epub 2018 Dec 3. PMID 30545649
- [Result] Billington J, Farrington G, Lampropoulou S, Lingwood J, Jones A, Ledson J, McDonnell K, Duirs N, Humphreys AL. A comparative study of cognitive behavioural therapy and shared reading for chronic pain. Med Humanit. 2017 Sep;43(3):155-165. doi: 10.1136/medhum-2016-011047. Epub 2016 Dec 9. PMID 27941097